CLINICAL TRIAL: NCT01053234
Title: Effects of Standardised Meals on Postprandial Coagulation Activation in Patients With Type 2 Diabetes Treated With Two Different Insulin Regimens
Brief Title: Different Insulin Regimens and Postprandial Coagulation Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Ribe County Hospital (Other); Novo Nordisk A/S (Industry)
Responsible Party: Chief physician, Ph.D Jeppe Gram, Department of Medicine, Hospital of South West Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRS 2006-1032
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes; Cardiovascular Risk; Hemostasis; Inflammation; Endothelial Function
Keywords: Hyperglycaemia; Postprandial; Type 2 diabetes; Cardiovascular risk markers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin aspart (Experimental)
  Interventions: Dietary Supplement: Standardised meals
- NPH insulin (Experimental)
  Interventions: Dietary Supplement: Standardised meals

INTERVENTIONS:
Dietary Supplement: Standardised meals

SUMMARY:
The purpose of this study in patients with type 2 diabetes was to investigate the acute effect of postprandial blood glucose levels modified by two different insulin treatment regimens on coagulation activation, inflammation and endothelial cell function. The investigators hypothesized that the rapid-acting insulin analogue aspart has a beneficial postprandial effect on coagulation, endothelial dysfunction and inflammation compared with the intermediate-acting insulin NPH due to its ability to lower postprandial glycaemia.

ELIGIBILITY:
Inclusion Criteria:

* age 30-75 years
* BMI > 25 kg/m2
* type 2 diabetes for more than 4 years
* pharmacological anti-diabetic treatment with insulin NPH at bedtime or insulin aspart at meals for more than 24 months
* metformin with stable dose >1000 mg/d for more than 12 weeks
* acetylsalicylic acid (75 mg/d) for more than 2 weeks
* no other anti-diabetic treatment 3 month previously
* HbA1c<8.5% at recruitment.

Exclusion Criteria:

* creatinine > 120 µmol/l
* ALAT /ASAT > 2.5 x upper reference limit
* use of anticoagulants within 1 month previously
* any changes in dose of statins within 1 month previously
* night work
* present or planned pregnancy
* mental sickness or alcohol abuse
* clinically relevant major organ or systemic illness
* uncontrolled hypertension >180/110 mmHg
* steroid treatment
* known or suspected allergy to trial medications.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Prothrombin fragment 1+2 | 7.40; 9.30; 11.30; 13.30; 15.30

SECONDARY OUTCOMES:
C-reactive protein | 7.40; 9.30; 11.30; 13.30; 15.30

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe Gram, Ph.D, Principal Investigator — Department of Medicine, Hospital of South West Denmark
Locations (1):
- Hospital of South West Denmark, Esbjerg, Denmark